CLINICAL TRIAL: NCT00841035
Title: University of Alabama at Birmingham(UAB 0808), A Phase II Study of Short-course Preoperative Erlotinib Followed by Post-operative Erlotinib-gemcitabine in Patients With Resectable Pancreatic Adenocarcinoma
Brief Title: 7 Day's of Erlotinib Neo-adjuvant, Followed by Adjuvant Erlotinib-gemcitabine in Pancreatic Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor stopped due to slow enrollment
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Marty Heslin, Chief of section of Surgical Oncology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F080718006
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic; Cancer; Assay; Biomarkers
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eroltinib added to standard of care (Experimental): 150 mg of erlotinib for 7 days prior to surgery,then in the adjuvant stage the subject will receive 100mg of erlotinib and gemcitabine 1000mg/2 for 6 cycles
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: erlotinib — Preoperative dosing of 150 mg oral erlotinib for 7 days before surgery. followed by erlotinib 100 mg daily 6 month/6 chemotherapy cycles. Gemcitabine 1000 m2 weekly after surgery for 6 cycles.
  Other Names: Tarceva

SUMMARY:
1.1 Primary Objective

To evaluate the effects of short course preoperative erlotinib treatment in a panel of predictive biomarkers from a group of patients who undergo resection of pancreatic adenocarcinoma with curative intent.

1.2 Secondary Objectives

1.2.1 To analyze the effects of short course preoperative erlotinib treatment followed by postoperative erlotinib-gemcitabine therapy in the disease-free survival of patients who undergo curative intent resection of pancreatic adenocarcinoma.

1.2.2 To evaluate secondary endpoints of disease response such as duration of overall survival and patterns of recurrence for patients with resectable pancreatic cancer who undergo this treatment regimen.

1.2.3 To evaluate the plasma pharmacokinetics of erlotinib in pancreatic cancer patients both in the preoperative and postoperative setting, and to explore correlations between plasma and tumor erlotinib concentrations.

1.2.4 To develop a clinically relevant predictive assay of response to erlotinib based on selected biomarkers in endoscopic ultrasound-fine needle aspiration (EUS-FNA) specimens when it can be obtained at the time of pancreatic cancer diagnosis in chemotherapy-naive patients.

DETAILED DESCRIPTION:
Our current clinical trial proposal includes a short course of pre-operative, single agent erlotinib followed by post-operative erlotinib-gemcitabine in a neo-adjuvant/adjuvant approach to the treatment of patients with resectable pancreatic adenocarcinoma. The short course pre-operative erlotinib treatment serves two objectives: 1) erlotinib, through its cytostatic effects, may hinder the ability of tumor cells to metastasize at the time of surgical resection with minimal toxic effects and no delay in surgical treatment; 2) the true effects of erlotinib on potential determinants of response can be best assayed on the pancreatic cancer itself since no other model can better resemble the patients authentic tumor microenvironment. The post-operative treatment component of the protocol attempts to improve the demonstrated effects of gemcitabine by adding erlotinib in the adjuvant setting, a drug combination that, as mentioned, has already been proven to be advantageous for patients with advanced pancreatic cancer.

Traditionally, chemotherapy for cancer has been conducted in an empiric fashion by first selecting a regimen based on clinical trial evidence and clinical parameters, and then by assessing the objective response to that regimen employing clinical and radiographic imaging means. This approach suffers from many disadvantages, most conspicuously the inability to select the better patient candidates prior to the initiation of therapy, thus sparing the risk and expense of ineffective treatment for patients who are unlikely to respond. Since pancreatic cancer expression of EGFR protein by itself is not predictive of therapeutic response, alternative methods of patient selection seem to be essential for the success of EGFR-targeted treatment. The understanding of EGFR molecular signaling has allowed the drug development process to shift from an empiric random screening approach to a more rational and mechanistic, target-directed approach. Among multiple attempts to identify molecular determinants of tumor cell sensitivity to EGFR inhibitors, there are two main paradigms that stand out: 1) activation of downstream pharmacodynamic effectors associated with response to the drug (i.e. phosphorylation of Akt or extracellular signal-regulated kinase (ERK); expression of c-fos), and 2) prediction of sensitivity based on a "static" analyte (detection of epidermal growth factor receptor (EGFR) sensitizing mutations; epithelial-mesenchymal transition profile). However, given the complexity of factors governing pancreatic cancer response to erlotinib, the biologic heterogeneity of malignant phenotype, and overall relatively low response rates, we believe that it is unlikely that analysis of a single biomarker will be useful for patient selection. A comprehensive analysis of a dynamic panel of biomarkers relevant to EGFR signaling and erlotinib mechanism of action seems more useful in that sense. Furthermore, the limited ability of pancreatic cancer tissue sampling often precludes biomarker correlation to assays worked out in xenograft models or in-vitro conditions.

The translational rationale of this proposal is therefore to develop predictive chemotherapy sensitivity-resistance assays (CSRA) for pancreas carcinoma patients treated with erlotinib and gemcitabine. This will represent a major advance, because the CSRA would enable prediction of clinical response prior to initiation of therapy.

ELIGIBILITY:
Inclusion Criteria:

.Histologic or cytologic confirmation of pancreatic ductal adenocarcinoma.

* Pancreatic cancer must be surgically resectable: a) no evidence of distant metastasis; b) clear fat plane around the celiac and superior mesenteric arteries; c) patent portal and superior mesenteric veins
* No evidence of post-resection distant metastasis
* Pathologic confirmation of R0/R1 status following surgical resection
* Age ≥ 19 years
* Male or female gender (not pregnant or lactating). If the subject is fertile, use of medically acceptable contraception will be required.
* Patient should be able to understand and offer signed written informed consent prior to study entry.
* No prior receipt of chemotherapy or radiotherapy
* Patients must demonstrate a Eastern Cooperative Oncology Group(ECOG) P.S. of 0 or 1
* End Organ function must be adequate meeting the below criteria at baseline:

White Blood Cell Count (WBC)> 3000/mm3, absolute neutrophil count(ANC)> 1500/mm3, Platelets>100,000mm3 Calculated creatinine clearance >50 ml/min, normal serum creatinine (mg/dL) (if calculated Crcl <50 ml/min, Crcl should measured and be > 50 ml/min) Bilirubin <3.0 mg/dL (patients with obstructive jaundice require preoperative endoscopic biliary stenting if total bilirubin >3.0 mg/dl) prothrombin time(PT) /partial thromboplastin time(PTT) below the upper limit of normal

Exclusion Criteria:

* Diagnosis of active (treated in past 5 years) concomitant malignancy with exception of non-melanotic skin cancer
* Transplant patients or patients receiving immunosuppression
* Presence of an underlying disease state associated with active bleeding or a past medical history of coagulopathy
* New York Heart Association Class IV congestive heart failure
* Limited mental capacity or language skills to the extent simple instructions cannot be followed or information regarding adverse events cannot be provided
* History of non-compliance with prescribed medical care

Post-Operative Phase Inclusion

* No Evidence of Post-Resection Distant Metastasis
* Pathological confirmation of R0/R1 status following Surgical resection
* Patient must demonstrate a post-operative performance status of 0 or 1.
* End Organ function must be adequate, meeting the below criteria at baseline:

  1. WBC > 3000/mm³,ANC > 1500/mm³, Platelets > 100,000 mm³
  2. Calculated Creatinine Clearance > 50 ml/min,Serum Creatinine < 1.5 mg/dl
  3. Bilirubin < 3.0 mg/dl; aspartate aminotransferase(AST) and alanine aminotransferase (ALT) < 3 x normal value
  4. PT/PTT/international normalized ratio(INR) within normal Limits.

     -

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Arnoletti, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham,Comprehensive Cancer Center, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Eroltinib Added to Standard of Care: 150 mg of erlotinib for 7 days prior to surgery,then in the adjuvant stage the subject will receive 100mg of erlotinib and gemcitabine 1000mg/2 for 6 cycles
  erlotinib : Preoperative dosing of 150 mg oral erlotinib for 7 days before surgery. followed by erlotinib-gemcitabine after surgery for 6 cycles.
Period: Phase 1 Overall Study
Arm/Group | Eroltinib Added to Standard of Care
Started | 19 (2 phase enrollment,1st phase enrolled with cancer by fine needle aspiration in endoscopic ultrasound)
Completed | 6
Not Completed | 13
Not completed — Physician Decision | 13
Period: Phase 2 of Overall Study
Arm/Group | Eroltinib Added to Standard of Care
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eroltinib Added to Standard of Care
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Secondary Outcome: The Secondary Objectives Include Analysis of Recurrence-free and Overall Survival and the Development of a Predictive Assay for Response to Erlotinib Based on Selected Bio-markers in Endoscopic Ultrasound-Fine-needle Aspiration Specimens.
Description: The measurement was to be the average length of time before recurrence of disease and the overall survival time. As well as time from recurrence to death in subjects.This time will be measure in months till recurrence and them months to death.
Time Frame: End of the study
Population: Due to the closure of the study before this endpoint could be met, there are no subjects analyzed.
Arm/Group | Eroltinib Added to Standard of Care
Number analyzed (Participants) | 0

2. Primary Outcome: Epidermal Growth Factor Receptor Signaling(EGFR) in the Presence of Pancreatic Tumor Related to the Mechanism to Erlotinib.
Description: It was our belief that we would need a comprehensive analysis of a dynamic panel of biomarkers relevant to EGFR signaling as well as the erlotinib mechanism of action it seems more useful in that sense. Furthermore,the ability limited of pancreatic cancer tissue sampling precluded biomarker correlation assays.These could not be worked out in either a xenograft model or in in-vitro conditions.
Time Frame: During the trial only
Arm/Group | Eroltinib Added to Standard of Care
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline to 36 month or subject death.
Arm/Group | Eroltinib Added to Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eroltinib Added to Standard of Care (N=19)
Chest Pain (Cardiac disorders) | 1 (1) — Subject had long standing history of cardiac disease and developed some chest pain after starting 7 days of erlotinib

LIMITATIONS AND CAVEATS:
Early termination by sponsor and No good clinical data was analyzed to the early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No